CLINICAL TRIAL: NCT05337241
Title: Saline Enhanced Radiofrequency (SERF) Needle Ablation for Refractory VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thermedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-90001
Record Dates: First submitted 2022-03-21; First posted 2022-04-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-08

CONDITIONS: Refractory Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Subjects with recurrent, SMVT refractory to drug therapy and conventional catheter ablation who are not eligible for, or will not likely benefit from repeat endocardial ablation using an approved catheter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm treatment (Experimental): All subjects meeting inclusion/exclusion criteria and successfully consented will be treated with the study device.
  Interventions: Device: Saline Enhanced Radiofrequency (SERF) Ablation

INTERVENTIONS:
Device: Saline Enhanced Radiofrequency (SERF) Ablation — The Durablate intramural needle catheter delivers heated saline to target tissue in the left ventricle to target mid-myocardial and epicardial VT substrates
  Other Names: Intramural Needle Ablation

SUMMARY:
The Thermedical Ablation System and Durablate catheter is indicated for use in patients with recurrent, sustained, monomorphic ventricular tachycardia (SMVT) refractory to drug therapy and conventional (approved) catheter ablation.

Subjects with recurrent, SMVT refractory to drug therapy and conventional catheter ablation who are not eligible for, or will not likely benefit from repeat endocardial ablation using an approved catheter.

DETAILED DESCRIPTION:
This is a staged, non-randomized, open-label, single group, interventional study to be conducted at up to 25 investigational sites to evaluate the safety and efficacy of the Thermedical Ablation System with the Durablate Ablation Catheter (investigational device) in subjects with recurrent, sustained, monomorphic ventricular tachycardia (VT) refractory to drug therapy and conventional catheter ablation.

Subjects will be consented (enrolled) and screened prior to the study ablation procedure. 154 subjects will have a study ablation procedure with the investigational device. Follow-up will occur at 7 days, 30 days, 3 months and 6 months.

The single arm design of the proposed study reflects the nature of the study population. The Thermedical Ablation System was designated as a Breakthrough technology in part because no currently approved device specifically treats this refractory patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has structural heart disease
2. Subject has recurrent symptomatic sustained (> 30 seconds) monomorphic ventricular tachycardia (MMVT) within 180 days prior to planned study ablation that meets the following criteria:

   1. At least 3 episodes of the MMVT have been treated with ATP and/or shock, OR at least 2 episodes were treated with shock AND
   2. Documentation of the presumed recurrent MMVT was treated with prior catheter ablation AND
   3. Occurred despite treatment with at least one Class III antiarrhythmic after last ablation or treatment with a Class III antiarrhythmic is not tolerated or is contraindicated AND
   4. VT has recurred despite VT ablation at one of the investigational centers UORU the investigator documents the reason that the subject is unlikely to benefit from a repeat ablation using a conventional, approved catheter.
3. Subject is at least 18 years old
4. Subject has an implantable cardioverter-defibrillator (ICD) with a full 6-month (prior to planned study ablation) ICD interrogation history documenting incidences of VT
5. Subject is able to provide informed consent

Exclusion Criteria:

1. Idiopathic VT (VT occurring in subjects without structural heart disease [including the absence of LGE on MRI, if performed], metabolic abnormalities or long QT syndrome)
2. Suspected area of ablation of target clinical VT includes aortic root, aortic cusp or any area outside left ventricle except the ventricular septum
3. Subject with a prior ablation within 4 weeks of planned study ablation
4. Subject's VT is not amenable to treatment with the study device at the time of mapping for the study ablation
5. Only PVCs are induced during mapping for the study ablation
6. No clinical VT induced during mapping for the study ablation
7. Planned use of a non-study ablation catheter
8. Subject has an LVEF < 20% reported on pre-ablation imaging (CT, MRI or echocardiogram within 48 hours of the study procedure)
9. Subject with evidence of any right- or left-sided (including left atrium, left atrial appendage and left ventricle) intracardiac thrombus OR pericardial effusion (except chronic trivial) reported on required pre-ablation imaging (CT, MRI, or echocardiography) or seen on required procedural intracardiac echocardiography (ICE) prior to study ablation catheter insertion.
10. Subjects with atrial fibrillation/flutter (paroxysmal, persistent, or permanent) without uninterrupted anticoagulation for at least 3 weeks immediately prior to the date of ablation procedure. (Interruption of anticoagulation in the day(s) just prior to ablation will be left to physician decision based upon subject's risk of stroke, anticoagulation agent, renal status, and bleed/embolic risk status with recommendation to consider bridging for high-risk subjects.
11. Subjects with NYHA Class IV heart failure
12. Renal dysfunction with eGFR <30 ml/min/1.73mP2
13. Subject with known coagulopathy or other condition likely to increase risk of periprocedural bleeding
14. Subject with known coagulopathy or other condition likely to increase risk of a thrombotic event
15. Subject with a mechanical aortic valve, mechanical mitral valve, or MitraClip
16. Subject with flail mitral leaflet or severe aortic stenosis
17. Subject with LAA occlusion device
18. Subject with a congenital heart defect except patent foramen ovale (PFO)
19. Subject with suspected life expectancy of less than 1 year
20. Subject with myocardial infarction (MI) or unstable angina (UA) within previous 90 days
21. Subject with cardiac surgery or percutaneous coronary intervention (PCI) within previous 90 days
22. Subject with known untreated significant ischemic coronary artery disease, acute illness (unrelated to VT or its origin) or active systemic infection.
23. Subject with left ventricular assist device planned or required for the procedure
24. Females who are or may potentially be pregnant (must be post-menopausal or have a negative pregnancy test)
25. Allergy or contraindications to the medications/agents used during a standard ablation/EP intervention including heparin and ionic contrast media
26. Contraindication to cardiac CT
27. Subject concurrently enrolled in any other investigational drug or device study that the investigator deems would interfere with study results
28. Subject with a condition (including a chronic illness) or circumstance that the investigator feels puts the subject at an unacceptable risk for participation in the study or may interfere with quality data collection or study results
29. Subject is not willing or is unable to participate in all study procedures and follow-up requirements

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-08-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy (Acute Interim) | At end of ablation procedure (ablation procedure occurs on a single day)
  Percentage of target clinical VTs that are non-inducible at end of the study ablation procedure (if PES performed at procedure conclusion)
Primary Efficacy (Long Term) | 6 month post ablation
  Percentage of subjects who are free from recurrent monomorphic VT

SECONDARY OUTCOMES:
Primary Safety | 7 days from intervention
  Per subject composite of cardiovascular-related and procedure-related major complications through 7 days post-study ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Curley, PhD, Study Director — Thermedical, Inc.
Locations (7):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Healthcare, Salt Lake City, Utah
- Canada (2):
  - Montreal Heart Institute - Institut de Cardiologie de Montréal, Montreal, Quebec
  - Quebec Heart and Lung Institute - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified and protected according to HIPAA